CLINICAL TRIAL: NCT06796738
Title: Advancing Cervical Cancer Screening Through the Emergency Department
Brief Title: Advancing Cervical Cancer Screening Through the Emergency Department - IIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, David Adler, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Study 00010129
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancers; HPV
Keywords: HPV; Cervical Cancer; Cancer Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention Arm - testing (Other): Participants in this arm will be provided the opportunity to self- sample for HPV during their ED visit. Participants will be (1) briefly instructed by the study staff on how to self-sample using a defined instructional script written at an elementary reading level, (2) provided with a packaged swab and vial of transport media, and (3) invited to self- sample privately in their ED room or in one of the private ED restrooms.
  Interventions: Diagnostic Test: HPV testing

INTERVENTIONS:
Diagnostic Test: HPV testing — This study will use the Roche Cobas® 8800 system for HPV testing. The Roche Cobas HPV test is a PCR test that detects 14 hrHPV types and specifically identifies types 16 and 18.

SUMMARY:
Cervical cancer screening in the Emergency Department

DETAILED DESCRIPTION:
This will be an effort to deploy HPV self-sampling among Emergency Department patients. Emergency Department patients, in the US and worldwide, are disproportionally under-screened for cervical cancer relative to the general population.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women and transgender/non-binary individuals with a cervix,
* Age 25-65,
* Able to demonstrate decisional capacity to participate.

Exclusion Criteria:

* Past hysterectomy with cervical removal,
* Known infection with HIV (as screening recommendations for people with HIV differ from the general population),
* Non-English speaking.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women and transgender/non-binary individuals with a cervix.
Enrollment: 200 (Actual)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of Cervical Cancer Screening | 150 days post initial intervention
  All intervention participants will receive a follow-up call at 150 days to assess uptake of any cervical cancer screening and for completion of the cervical cancer screening process. "Any cervical cancer screening" is defined as uptake of any aspect of the cervical cancer screening process, including self-sampling and/or clinic-based screening. "Completion of the cervical cancer screening process" is defined as completion of recommended clinic-based screening (including colposcopy if HPV 16/18+ or indicated).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided